CLINICAL TRIAL: NCT06616090
Title: Investigating the Effectiveness of Nurse Implemented Attachment-Based Maternal Sensitivity Program in Primary Family Health Care Services
Brief Title: Nurse Implemented Infant-Mother Attachment Security Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sabanci University (Other)
Responsible Party: Principal Investigator, Feyza Corapcı, Professor of Psychology, Sabanci University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 123K416
Record Dates: First submitted 2023-12-01; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2023-12

CONDITIONS: Nurse's Role; Infant Development; Maternal Behavior
Keywords: attachment-based program; maternal sensitivity; attachment security; nurse-based; primary healthcare

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be conducted. The sample will consist of 120 mothers with 9- to 12-month-old babies from Family Health Centers (FHC) in Istanbul. FHCs will be randomly assigned to intervention and control conditions so that mother-infant dyads will be divided into intervention (N = 60) and control (N = 60) groups. A comprehensive training will be provided to intervention nurses. Mother-infant dyads in the intervention group will receive the regulare well child check up procedures along with the attachment-based intervention modules, following the pretest measurements. Mother-infant dyads in the control group will receive the routine well-child check up procedures. Changes in maternal sensitivity and infant attachment security from pre- to posttest will be compared across two groups measures. Control mothers will receive a condensed form of the intervention after the follow up assessments.
Who Masked: Outcomes Assessor
Masking Description: The assessment team will be blind to the treatment condition of the mothers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nurse implementation (Experimental): This arm will receive nurse implemented attachment-based parenting modules in addition to routine well-child check up
  Interventions: Behavioral: Nurse Implemented Infant-Mother Attachment Security Program
- No intervention (No Intervention): This arm will receive routine well-child check up

INTERVENTIONS:
Behavioral: Nurse Implemented Infant-Mother Attachment Security Program — The intervention will draw on video-feedback of mother-infant interactions during the well-child visit. Nurses will videotape the dyad during routine visit in the Family Health Center and show short clips to mothers during the session in order to provide mother positive feedback on their sensitive caregiving. Additionaly, intervention mothers will be exposed to the reminders (e.g., pictures, posters, short film screenings) reflecting maternal sensitivity and secure attachment in the waiting rooms of the intervention Family Health Centers.
  Arms: Nurse implementation

SUMMARY:
This study focuses on adapting and evaluating an attachment-based intervention program implemented by nurses in Family Health Centers (FHCs) in Turkey. The program aims to enhance parental sensitivity and infant-mother attachment security. Evidence suggests that such programs, developed in Western countries, effectively improve parenting behaviors and attachment quality. Despite the positive effects of similar programs in Turkey, their integration into primary healthcare for wider public benefit remains unexplored. The project will develop an intervention protocol based on effective methods from previous attachment-based programs into routine childcare visits at FHCs. A randomized controlled trial involving 120 mothers with 9- to 12-month-old babies in Istanbul will be recruited. FHCs will be randomly assigned to intervention and control groups, with 60 mother-infant dyads in each condition. Nurses will deliver the program during childcare visits at 9, 12, 15, and 18 months. Intervention FHCs will also use reminders like posters and short films in the waiting rooms to reinforce the concepts. Effectiveness will be evaluated through pretest, posttest, and follow-up home visits using observational and self-report measures on attachment security, maternal sensitivity, as well as maternal psychological characteristics, along with infant socioemotional measures. Upon completion of the project, control FHC nurses will receive training to deliver a condensed version of the program.

DETAILED DESCRIPTION:
This study aims to adapt and evaluate the effectiveness of an attachment-based, protective-preventive intervention program implemented by nurses in Family Health Centers (FHC) that routinely follow up infants' health. Attachment-based parenting intervention programs have been developed and implemented in Western countries given that parental sensitivity and secure attachment relationship in the early years are critical precursors of psychological resilience. These evidence-based programs have been widely shown to reinforce responsive parenting behaviors and improve attachment quality. A few attachment-based programs have been adopted in Turkey with documented positive effects. However, adaptations of such programs within the primary healthcare services that actively reach families have yet to be conducted to evaluate their potential widespread use for public benefit. In this proposed project, effective application methods of attachment-based programs identified in previous studies, will be integrated to the current well-child care visits in FHCs. It is expected that this program will positively affect maternal sensitivity, caregiving competence, positive discipline methods, mother-child attachment security, and reduce child problem behaviors (e.g., internalizing and externalizing problems). It is also expected that the program effectiveness will be more robust among mothers from socioeconomically disadvantaged families, those with initially low levels of sensitivity, and anxious attachment pattern. To test these expectations with a randomized controlled trial, 120 mothers with 9-month-old babies from FHCs in Istanbul will participate. Selected FHCs will be randomly assigned to intervention and control conditions. Mother-infant dyads will be divided into intervention (N = 60) and control (N = 60) groups. Following a comprehensive training, nurses will apply five modules with sensitivity and positive discipline themes, including a booster module, to the mother-infant dyads during well-child care visits at the 9th, 12th, 13th, 14th and 15th months following the pretest measurements. The application will draw on nurses' positive feedback to mothers utilizing short video recordings and in-the-moment mother-baby interactions consistent with each module theme. Additionaly, mothers will be exposed to the reminders (e.g., pictures, posters, short film screenings) reflecting maternal sensitivity and secure attachment in the waiting rooms of the intervention FHCs. The proposed project will be carried out by experts from psychology with research and experience in attachment-based intervention in collaboration with the experts working in family medicine, nursing, and primary healthcare. To examine program effectiveness, pretest, posttest, and follow-up measurements will occur at pre-defined times through home visits to mothers. Data on mother and infant demographics and psychological characteristics will be collected using multimethod measurement in line with the program goals. Thus, maternal sensitivity level will be assessed using the Ainsworth Sensitivity Scale and Maternal Sensitivity Q-Sort, and the mother-infant attachment quality will be assessed using the short form of the Attachment Q-Sort. Besides observation, mother-reported sensitivity and attitudes towards discipline, caregiving competence, mental processes underlying child's emotions and behaviors, and psychological characteristics (e.g., adult attachment pattern, depressive symptoms) will be evaluated with widely used measurement tools. Finally, infant development and temperament will be assessed via mother report. Following the intervention program, training will also be given to nurses in the control FHCs, who will deliver a condensed maternal sensitivity program to control mothers. The program will be disseminated to relevant experts and institutions, including the priority stakeholders in the family primary healthcare system. If the program's effectiveness is demonstrated, special efforts will be made to scale-up the program. Given that attachment-based early intervention programs positively affect child development throughout life, improve the family environment and social relations and reduce public expenditure on health problems in the long run, the proposed program is expected to create a similar impact in Turkey and lead to positive psychosocial change.

ELIGIBILITY:
Inclusion Criteria:

* mothers with 9- to 12-month infants
* having a normally developing infant.

Exclusion Criteria:

* mothers with infants who have a chronic pediatric health problem
* mother with infants whose developmental problems are detected during routine evaluations
* mothers with temporary protection status (i.e., immigrants) due to potential communication problems
* if the mother is not the primary caregiver

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Maternal sensitivity 1 | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  The Ainsworth Sensitivity Scale (Ainsworth et al., 1978) will be used to assess maternal global sensitivity. The scale ranges from 1 to 7, with higher scores meaning higher maternal sensitivity
Maternal sensitivity 2 | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  Maternal Behavior Q-set will be used to assess maternal global sensitivity. The score ranges from -1 (extremely insensitive) to +1 (extremely sensitive).
Attachment Security | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  Attachment Q-sort will be used to assess the security of infant attachment. Scores range from -1 (high levels of attachment insecurity) to +1 (high levels of attachment security)
Maternal Sensitive Discipline | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  Maternal Attitudes toward Sensitivity and Sensitive Discipline Scale will be used. The scale score ranges from 1 to 6. Higher scores characterize mothers with more sensitive attitudes towards sensitive care and discipline.
Infant Socio-Emotional Development | Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  The Problem Behaviors Subscale of the Brief Infant Toddler Socioemotional Assessment scale will be used to measure age-relevant developmental difficulties in young children. Scores range from 0 to 62, with higher scores characterizing children with more frequent behavioral and emotional problems.

SECONDARY OUTCOMES:
Maternal Reflective Functioning | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  Mothers' ability to mentalize their children will be measured with the Pre-Mentalizing Modes of the Parental Reflective Functioning Questionnaire. Scores range from 1 to 7. Higher scores indicate higher levels of impairment in parental reflective functioning such as parents' lack of acknowledgement for the child's subjective world.
Maternal Attachment Representation | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  The short form of the Experiences in Close Relationships questionnaire will be used to measure mothers' attachment anxiety and avoidance. Scores for attachment anxiety range from 1 to 6, with higher scores indicating higher levels of attachment anxiety in mothers. Scores for attachment avoidance range from 1 to 6, with higher scores indicating higher levels of attachment avoidance in mothers.
Maternal Efficacy in Parenting | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  Mothers' sense of competence in dealing with infant care and parenting will be measured with a subscale from the Parenting Stress Index. The scores range from 1 to 6, with higher scores higher perceived competence in parenting.
Maternal depression | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  Maternal psychological well being will be measured by using the Edinburgh Postpartum Depression scale. The scores range from 0 to 30 with higher scores indicating higher levels of maternal depression
General Parenting Practices | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  Maternal warmth, cognitive stimulation and general discipline practices will be measured with the Comprehensive Early Childhood Parenting Questionnaire. Scores range from 1 to 6 with higher scores indicating better quality caregiving.
Marital Conflict | Pretest: 1 month before the intervention begins when infants are 8 months old. Posttest: Immediately after the intervention concludes, when infants are 18 months old. Follow-up: 2 months after the the intervention ends, when infants are 20 months old
  Spousal disagreement over child rearing will be measured with the O'Leary-Porter scale of marital conflict. Scores range from 1 to 4, with higher scores indicating more frequent spousal disagreement in front of the child.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Çorapçı, PhD, Principal Investigator — Sabanci University
Locations (1):
- Sabanci University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Open science guidelines will be followed
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available in 2027